CLINICAL TRIAL: NCT07131397
Title: The Effect of Inspiratory Muscle Training on Inspiratory Strength in People With Gastroesophageal Reflux Disease.
Brief Title: The Effect of Inspiratory Muscle Training in People With Gastroesophageal Reflux Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Responsible Party: Principal Investigator, IRINI PATSAKI, Assistant professor, University of West Attica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10545
Record Dates: First submitted 2025-08-10; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Gastro Esophageal Reflux
Keywords: Inspiratory Muscle Training; Gastroesophageal Reflux Disease; Antireflux valve; Maximal Inspiratory Pressure
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory Muscle Training (Experimental): Inspiratory muscle training will be applied with the K5 Power Breath trainer. The exercise will be performed by applying resistance at 40% of the maximum inspiratory pressure (1 set of 30 repetitions 30 breaths per session). Each week there will be a gradual increase in resistance by 10% of the initial maximum inspiratory pressure.
  Interventions: Device: Inspiratory Muscle Traing
- Control (Sham Comparator): Inspiratory muscle training will be applied with a constant resistance load of 7cmH20.
  Interventions: Device: Sham Inspiratory Muscle Training

INTERVENTIONS:
Device: Inspiratory Muscle Traing — IMT will be performed by applying resistance at 40% of the maximum inspiratory pressure (1 set of 30 repetitions 30 breaths per session). Each week there will be a gradual increase in resistance by 10% of the initial maximum inspiratory pressure.
  Arms: Inspiratory Muscle Training
Device: Sham Inspiratory Muscle Training — Inspiratory muscle training will be applied with a constant resistance load of 7cmH20
  Arms: Control

SUMMARY:
The present Randomized Control Trial will be a single centric, two arm parallel equivalence randomized controlled. Participants will be assigned to either the Inspiratory MuscleTraining (IMT) group (investigation) or to Sham IMT group (control). The assessment times were three (3) before the start of the program (baseline-T1), immediately after the 3 months of the main exercise program (end of the main program-T2) and 6 months after (end of follow up-T3).

The measurements included: A. By measuring the Maximum Inspiratory Pressure (MIP) (Micro RPM) B. By measuring the Maximum Dynamic Inspiratory Pressure s-index (Powerbrethe K5)

The following instruments were included in the secondary outcome measures:

* Recurrent Gastroesophageal Reflux Disease Questionnaire (measurement of symptom frequency-RDQ Questionaire).
* Gastroesophageal Reflux Disease-Related Quality of Life Questionnaire (Quality of Life Measure-Reflux Qual short form questionnaire).

DETAILED DESCRIPTION:
Background: Gastroesophageal reflux disease (GERD) is multifactorial and affects an increasing number of people. Its main cause is found in the antireflux valve mechanism of the gastroesophageal junction. This consists of two sphincters, the lower oesophageal and the diaphragmatic. The disease has been related to diaphragm dysfunction, either due to the de-coordination of the diaphragms' contractility or due to decreased strength. This study was designed to evaluate the effect of inspiratory muscle training on inspiratory strength in people with gastroesophageal reflux disease.

Objective: To evaluate the effect of a IMT program in maximal inspiratory pressure, maximal dynamic inspiratory pressure, gerd symptoms and quality of life in GERD patients.

Methods: Adults with diagnosed gastroesophageal reflux disease (n=30) or had a score of more than 8 on the Gastroesophageal Reflux Disease Questionnaire will be recruited from invitations that will be made through the social media. The volunteers who meet the inclusion criteria will be randomly allocated to two groups: (a) the experimental group (n = 15) that will receive 36 sessions inspiratory muscle training with tapered flow resistive loading at 40% of maximum inspiratory pressure. Each week there will be a gradual increase in resistance by 10% of the initial maximum inspiratory pressure. (b) Τhe control group (n = 15) that will receive 36 sessions inspiratory muscle training with a constant resistance load of 7cmH20 (sham group). Both groups will perform 3 sessions per week (1 set of 30 repetitions). Measurements will occur at three time points: before the initiation of treatment sessions (week 0), three months from the beginning of the trial (week 36) and 6 months after the end of the program. The main outcomes will be the maximal respiratory pressures (digital pressure manometer), maximal dynamic inspiratory pressure (tapered flow resistance device) with secondary outcomes the gerd symptoms (gerd-q questionnaire) and quality of life (Reflux Qual short form questionnaire).

Anticipated Results: IMT is expected to increased Mip, S-Index, improve Reflux Symptoms and quality of life, mitigate the impact of gerd in the participants' health and daily life compared to standard care.

Conclusion: This trial will provide novel insights into IMT's role in symptoms prevention for GERD patients, addressing a critical gap in holistic disease management.

ELIGIBILITY:
Inclusion Criteria: people diagnosed with GERD or had a score of more than 8 on the Gastroesophageal Reflux Disease Questionnaire

Exclusion Criteria: systemic connective tissue diseases, mental disorders, stomach or duodenal surgery, tuberculosis, pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure | the start of the program (baseline-T1), immediately after the 3 months of the main exercise program (end of the main program-T2) and 6 months after (end of follow up-T3)

SECONDARY OUTCOMES:
Maximum Dynamic Inspiratory Pressure s-index | the start of the program (baseline-T1), immediately after the 3 months of the main exercise program (end of the main program-T2) and 6 months after (end of follow up-T3)
Gastroesophageal Reflux Disease Questionnaire | Before the start of the program (baseline-T1), immediately after the 3 months of the main exercise program (end of the main program-T2) and 6 months after (end of follow up-T3).
Gastroesophageal Reflux Disease-Related Quality of Life Questionnaire | Before the start of the program (baseline-T1), immediately after the 3 months of the main exercise program (end of the main program-T2) and 6 months after (end of follow up-T3).

CONTACTS AND LOCATIONS:
Locations (1):
- University of West Attica, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No